CLINICAL TRIAL: NCT01342640
Title: A Single Arm, Open Label, Multicenter Phase IIIb/IV Clinical Trial to Assess the Efficacy, Safety and Tolerability of Monthly Administration of C.E.R.A. for the Treatment of Not on Dialysis Chronic Renal Anemia Not Currently Treated With ESA
Brief Title: A Study of Mircera (C.E.R.A.) in Patients With Pre-Dialysis Chronic Renal Anemia
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ML25300
Record Dates: First submitted 2011-04-20; First posted 2011-04-27 (Estimated); Results first posted 2015-10-26 (Estimated); Last update posted 2017-07-12 (Actual); Status verified 2017-06

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia | interventions — continuous erythropoietin receptor activator

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental)
  Interventions: Drug: methoxy polyethylene glycol-epoetin beta [Mircera]

INTERVENTIONS:
Drug: methoxy polyethylene glycol-epoetin beta [Mircera] — Recommended starting dose 1.2 micrograms/kg subcutaneously every 4 weeks (depending on patient's weight). Dose adjustment may be required in the event of inadequate or excessive treatment response.

SUMMARY:
This single arm, open label, multicenter study will evaluate the safety and change in hemoglobin levels of Mircera (C.E.R.A.; methoxy polyethylene glycol-epoetin beta) in patients with chronic renal anemia who are not on dialysis. Patients will receive as a recommended starting dose 1.2 micrograms of Mircera subcutaneously every 4 weeks. The starting dose is dependent on the patient's weight. Dose adjustment may be required due to inadequate or excessive treatment response. The anticipated time on study treatment is 28 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, age >/=18 years
* Diagnosis of chronic renal anemia
* Not on dialysis
* Hemoglobin concentration <10 g/dl
* No erythropoiesis stimulating agent (ESA) therapy during the 3 months before study start
* Estimated glomerular filtration rate (EGFR) <60 ml/min and >/=20 ml/min
* Adequate iron status

Exclusion Criteria:

* Transfusion of red blood cells during the previous 2 months
* Poorly controlled hypertension
* Significant acute or chronic bleeding, e.g. gastrointestinal bleeding
* Active malignant disease (except non-melanoma skin cancer)
* Hemolysis
* Hemoglobinopathies, e.g. sickle-cell disease, thalassemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2011-07-18 (Actual); Primary Completion 2012-11-30 (Actual); Study Completion 2012-11-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (5):
- Egypt (5):
  - Mansoura Kidney Center; Nephrology, Al Mansurah
  - Alexandria University; Endocrinology Department, Alexandria
  - El Qahira Al Fatemeya Hospital, Cairo
  - Kasr El Ainy University Hospital; Endocrinology Department, Cairo
  - Nasser Institute, Cairo

RESULTS

PARTICIPANT FLOW:
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants received methoxy polyethylene glycol-epoetin beta (Mircera, Continuous Erythropoietin Receptor Activator [C.E.R.A]) at a starting dose of 1.2 micrograms per kilogram (mcg/kg) administered via subcutaneous (SC) injection every 4 weeks for 28 weeks. Doses were adjusted according to individual's hemoglobin (Hb) level.
Period: Overall Study
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Started | 70
Completed | 29
Not Completed | 41
Not completed — Adverse Event | 3
Not completed — Protocol Violation | 16
Not completed — Lost to Follow-up | 21
Not completed — Other | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: All participants who received at least 1 dose of methoxy polyethylene glycol-epoetin beta treatment and for whom at least 1 follow-up data was available.
Groups:
- Methoxy Polyethylene Glycol-Epoetin Beta: Participants received methoxy polyethylene glycol-epoetin beta at a starting dose of 1.2 mcg/kg administered via SC injection every 4 weeks for 28 weeks. Doses were adjusted according to individual's Hb level.
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.80 (16.68)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 25

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Hb Concentration at Week 20
Description: Per Protocol (PP) Population: All participants in the safety population (all enrolled participants) except participants with less than 3 recorded Hb values in Weeks 20 to 28; who missed methoxy polyethylene glycol-epoetin beta dose in Weeks 20 to 28; who withdrew before efficacy evaluation period (Weeks 20 to 28); and participants with inadequate iron status (defined as mean serum ferritin less than or equal to [≤] 100 nanogram per milliliter [ng/mL] or mean transferrin saturation [TSAT] ≤20% or mean hypochromic red blood cells [RBCs] greater than or equal to [≥] 10% during efficacy evaluation period [Weeks 20 to 28]).
Time Frame: Baseline (Week 0), Week 20
Population: PP Population. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome and n signifies those participants who were evaluable for specified time-point.
Measure: Mean (Standard Deviation); unit: Grams per deciliter (gm/dL)
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 53
Grams per deciliter (gm/dL)
  Baseline (n=53) | 8.820 (0.736)
  Change at Week 20 (n=35) | 1.440 (1.144)
Statistical Analysis 1: Comparison: Methoxy Polyethylene Glycol-Epoetin Beta; Change from baseline in mean Hb levels at Week 20 was analyzed using paired t-test; Test type: Superiority or Other; p < 0.0001, Paired t-test

2. Primary Outcome: Change From Baseline in Mean Hb Concentration at Week 24
Description: PP Population: All participants in the safety population (all enrolled participants) except participants with less than 3 recorded Hb values in Weeks 20 to 28; who missed methoxy polyethylene glycol-epoetin beta dose in Weeks 20 to 28; who withdrew before efficacy evaluation period (Weeks 20 to 28); and participants with inadequate iron status (defined as mean serum ferritin ≤ 100 ng/mL or TSAT ≤20% or mean hypochromic RBCs ≥ 10% during efficacy evaluation period [Weeks 20 to 28]).
Time Frame: Baseline (Week 0), Week 24
Population: PP Population. Here, number of participants analyzed (N) signifies those participants who were evaluable for this outcome.
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 32
gm/dL | 1.470 (1.236)
Statistical Analysis 1: Comparison: Methoxy Polyethylene Glycol-Epoetin Beta; Change from baseline in mean Hb levels at Week 24 was analyzed using paired t-test; Test type: Superiority or Other; p < .0001, Paired t-test

3. Primary Outcome: Change From Baseline in Mean Hb Concentration at Week 28
Description: as for outcome 2
Time Frame: Baseline (Week 0), Week 28
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: gm/dL
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Number analyzed (Participants) | 28
gm/dL | 1.680 (1.115)
Statistical Analysis 1: Comparison: Methoxy Polyethylene Glycol-Epoetin Beta; Change from baseline in mean Hb levels at Week 28 was analyzed using paired t-test; Test type: Superiority or Other; p < .0001, Paired t-test

ADVERSE EVENTS:
Time Frame: From screening up to 32 Weeks
Arm/Group | Methoxy Polyethylene Glycol-Epoetin Beta
Serious Adverse Events (participants affected / at risk) | 7/70
Other Adverse Events (participants affected / at risk) | 7/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=70)
Renal failure chronic (Renal and urinary disorders) | 1
Peripheral ischemia (Vascular disorders) | 1
Renal failure (Renal and urinary disorders) | 1
Pneumonia cytomegaloviral (Infections and infestations) | 1
Hemoglobin decreased (Investigations) | 1
Complications of transplanted kidney (Injury, poisoning and procedural complications) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methoxy Polyethylene Glycol-Epoetin Beta (N=70)
Urinary tract infection (Infections and infestations) | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.